CLINICAL TRIAL: NCT01593826
Title: Pharmacokinetic Study Comparing Two Budesonide/Formoterol Fumarate Dihydrate Device-metered Dry Powder Inhalers, Budesonide/Formoterol Easyhaler 320/9 Microg/Inhalation and Symbicort Turbuhaler Forte; a Randomised, Double-blind, Single Centre, Single Dose, Crossover Study in Healthy Subjects
Brief Title: Comparison of Absorption of Budesonide and Formoterol From Budesonide/Formoterol Easyhaler and Symbicort Turbuhaler
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3103010
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Charcoal; Budesonide; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Charcoal and Symbicort Turbuhaler (Active Comparator)
  Interventions: Drug: Charcoal and Symbicort Turbuhaler
- Symbicort Turbuhaler (Active Comparator)
  Interventions: Drug: Symbicort Turbuhaler forte
- Charcoal and Budesonide/formoterol Easyhaler (Experimental)
  Interventions: Drug: Charcoal and Budesonide/formoterol Easyhaler 320/9 microg
- Budesonide/formoterol Easyhaler (Experimental)
  Interventions: Drug: Budesonide/formoterol Easyhaler 320/9 microg

INTERVENTIONS:
Drug: Charcoal and Budesonide/formoterol Easyhaler 320/9 microg — 2 inhalations as a single dose
  Arms: Charcoal and Budesonide/formoterol Easyhaler
Drug: Charcoal and Symbicort Turbuhaler — 2 inhalations as a single dose
  Arms: Charcoal and Symbicort Turbuhaler
Drug: Budesonide/formoterol Easyhaler 320/9 microg — 2 inhalations as a single dose
  Arms: Budesonide/formoterol Easyhaler
Drug: Symbicort Turbuhaler forte — 2 inhalations as a single dose
  Arms: Symbicort Turbuhaler

SUMMARY:
The purpose of this study is to compare the test product Budesonide/formoterol Easyhaler with the marketed product Symbicort Turbuhaler in terms of the drug absorbed into the bloodstream.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females aged 18-60 years.
2. Normal weight, at least 50 kg.

Exclusion Criteria:

1. Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, GI, pulmonary, metabolic-endocrine, neurological or psychiatric disease.
2. Any clinically significant abnormal laboratory value or physical finding that may interfere with the interpretation of study results or constitute a health risk for the subject if he/she takes part in the study.
3. Any condition requiring regular concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during the study.
4. Known hypersensitivity to the active substance(s) or the excipient of the drug.
5. Pregnant or lactating females.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter Cmax of plasma budesonide concentration | within 12 h
Pharmacokinetic parameter Cmax of plasma formoterol concentration | within 24 h
Pharmacokinetic parameter AUCt of plasma budesonide concentration | Within 12 h
Pharmacokinetic parameter AUCt of plasma formoterol concentration | Within 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Leena Mattila, MD, PhD, Principal Investigator — Orion Corporation, Orion Pharma; Ulla Sairanen, MSc, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- Orion Pharma Clinical Pharmacology Unit, Espoo, Finland